CLINICAL TRIAL: NCT02678624
Title: Project Collabri. The Effects of a Danish Model of Collaborative Care for People With Anxiety in General Practice
Brief Title: Project Collabri for Treatment of Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2013-203-A
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety; Social Phobia; Panic Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment according to the Collabri model (Experimental): Participants in this group will recive treatment according to the Collabri model which is a Danish model for collaborative care between primary and secondary care for depression, social phobia, generalized anxiety and panic disorder
  Interventions: Other: Treatment according to the Collabri model
- Treatment as usual (No Intervention): Control group. Participants in this group will recive treatment as usual. This means that participants will recive treatment corresponding to what their GP normally would offer as treatment. E.g. this could be refferal to a psychologist or psychiatrist and/or medicine.

INTERVENTIONS:
Other: Treatment according to the Collabri model — The Collabri Model is a complex intervention and consists of a number of treatment modalities. The Collabri Model includes the following elements: A multi-professional approach to treatment including a care manager, scheduled monitoring and review, enhanced inter-professional communication and a structured treatment plan. It further integrates: Recruitment of staff with psychiatric experience, training of general practitioner and care manager, use of instruments for detection and follow-up, education and treatment of the patient, supervision from a psychiatric specialist, guided self-help, patient- and relative involvement and a stepped care approach to treatment where treatment is always commenced on the least invasive and least resource-demanding level.
  Arms: Treatment according to the Collabri model

SUMMARY:
The purpose of this study is to determine whether treatment of patients with anxiety according to the Collabri Model is more effective in reducing symptoms compared to treatment as usual (TAU)

DETAILED DESCRIPTION:
Background:

Depression and anxiety are common diseases often treated in general practice. However, there are obstacles for optimal treatment e.g. a lack of continuity in disease management, organized collaboration between primary and secondary care and access to psychotherapy. Previous collaborative care studies have shown significant improvements in treatment outcomes for patients with depression and anxiety in primary care; however studies have yet not been carried out in a Danish context. Thus, the Collabri-model for collaborative care for panic disorder, generalized anxiety, social phobia and depression has been developed. The model includes: a multi-professional approach to treatment including a care manager (e.g. a psychiatric nurse), enhanced inter-professional communication, scheduled monitoring and review and structured treatment plans.

Objective:

To investigate whether treatment according to the Collabri-model have an effect on symptoms for people with anxiety disorders.

Methods/design:

Three cluster-randomized, clinical trials are set up to investigate treatment according to the Collabri-model compared to treatment as usual for 364 patients diagnosed with panic disorder, generalized anxiety and social phobia respectively from general practices in the Capital Region of Denmark. For all studies, the primary outcome is anxiety symptoms measured with Beck Anxiety Inventory (BAI) at 6 months.

Results/discussion:

The results will contribute new knowledge on collaborative care for depression and anxiety disorders in Danish conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18+ years
* Danish speaking
* Diagnosis of current depression using the Mini International Neuropsychiatric Interview (MINI) (DSM IV) by researchers that have been trained in using MINI and according to the ICD-10 criteria or when diagnosed by GP after conference with a psychiatrist in Project Collabri
* The patient has given her/his written informed consent to participate in the trial at the described terms

Exclusion Criteria:

* High risk of suicide assessed in the Mini International Neuropsychiatric Interview (MINI) and/or by general practitioner
* Psychotic condition detected in the MINI and/or by general practitioner
* Patients with a diagnosis of dementia
* Pregnancy
* Alcohol or substance misuse that hinders the person participating in Collabri treatment as assessed by the practitioner or researcher at inclusion interview
* Patients that are in current psychological or psychiatric treatment due to anxiety or depression
* Patients with a pending disability pension case
* Patients who have been treated for anxiety or depression within the last 6 months
* For patients in the intervention group: Patients with depression who wants treatment cf. the Danish psychologist scheme and do not want the reference to the psychologist preceded by other treatment, cf. the Collabri model
* For patients in the intervention group: If the patient at the first point of contact with the general practitioner after inclusion by a research assistant is referred to treatment as a part of the secondary psychiatric care system.
* Patients who are assessed by the general practitioner as medically unstable making it impossible for the patient to adhere to treatment
* OCD, PTSD, bipolar affective disorder as assessed in the MINI and/or by the general practitioner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Degree of anxiety measured by the Beck Anxiety Inventory (BAI) | At 6 months follow up after baseline
  The measure is self-reported

SECONDARY OUTCOMES:
Degree of depression measured by the Beck Depression Inventory (BDI) | At 6 months follow up after baseline
  The measure is self-reported
Psychological stress measured with the Symptom Checklist (SCL-92) | At 6 months follow up after baseline
  The measure is self-reported
Functional impairment measured with the Global Assessment of Functioning (GAF-F split version) | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview

OTHER OUTCOMES:
Degree of anxiety measured by the Beck Anxiety Inventory (BAI) | At 15 months follow up after baseline
  The measure is self-reported
Degree of depression measured by the Beck Depression Inventory (BDI) | At 15 months follow up after baseline
  The measure is self-reported
Psychological stress measured with the Symptom Checklist (SCL-92) | At 15 months follow up after baseline
  The measure is self-reported
Functional impairment measured with the Global Assessment of Functioning (GAF-F split version) | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview
Quality of life measured with the WHO-5 scale | At 6 months follow up after baseline
  The measure is self-reported
Quality of life measured with the WHO-5 scale | At 15 months follow up after baseline
  The measure is self-reported
Personal and social performance measured with the Personal and Social Performance scale (PSP) | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview
Personal and social performance measured with the Personal and Social Performance scale (PSP) | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview
Side effects measured by the PRISE questionnaire | At 6 months follow up after baseline
  The measure is self-reported
Side effects measured by the PRISE questionnaire | At 15 months follow up after baseline
  The measure is self-reported
Health-related quality of life measured with the EQ-5D | At 6 months follow up after baseline
  The measure is self-reported
Health-related quality of life measured with the EQ-5D | At 15 months follow up after baseline
  The measure is self-reported
Functional impairment measured with Sheehan Disability Scale (SDS) | At 6 months follow up after baseline
  The measure is self-reported
Functional impairment measured with Sheehan Disability Scale (SDS) | At 15 months follow up after baseline
  The measure is self-reported
Sick leave | At 6 months follow up after baseline
  The measure is obtained from the Danish DREAM database
Sick leave | At 15 months follow up after baseline
  The measure is obtained from the Danish DREAM database
Self-efficacy measured with the subscale "Obtain Help from Community, Family, Friends" from the Chronic Disease Self-Efficacy Scale | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Obtain Help from Community, Family, Friends" from the Chronic Disease Self-Efficacy Scale | At 15 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Control/Manage Depression Scale" from the Chronic Disease Self-Efficacy Scale | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Control/Manage Depression Scale" from the Chronic Disease Self-Efficacy Scale | At 15 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Personal Control" from The Revised Illness Perception Questionnaire (IPQ-R) | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Personal Control" from The Revised Illness Perception Questionnaire (IPQ-R) | At 15 months follow up after baseline
  The measure is self-reported
Apathia | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview
Apathia | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD PhD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curth NK, Brinck-Claussen UO, Hjorthoj C, Davidsen AS, Mikkelsen JH, Lau ME, Lundsteen M, Csillag C, Christensen KS, Jakobsen M, Bojesen AB, Nordentoft M, Eplov LF. Collaborative care for depression and anxiety disorders: results and lessons learned from the Danish cluster-randomized Collabri trials. BMC Fam Pract. 2020 Nov 18;21(1):234. doi: 10.1186/s12875-020-01299-3. PMID 33203365
- [Derived] Curth NK, Brinck-Claussen UO, Davidsen AS, Lau ME, Lundsteen M, Mikkelsen JH, Csillag C, Hjorthoj C, Nordentoft M, Eplov LF. Collaborative care for panic disorder, generalised anxiety disorder and social phobia in general practice: study protocol for three cluster-randomised, superiority trials. Trials. 2017 Aug 16;18(1):382. doi: 10.1186/s13063-017-2120-3. PMID 28814317